CLINICAL TRIAL: NCT02665104
Title: Investigation of Blood Flow Velocity in the MCA and Oxygen Saturation of the Brain During Carotid Endarterectomy in Local Anesthesia in Patients With and Without Neurological Symptoms Using Transcranial Doppler (TCD) and INVOS Monitor
Brief Title: Middle Cerebral Artery Velocity and Oxygen Saturation of the Brain During Carotid Endarterectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, assistant professor anesthesiologist and intensive care specialist, University of Debrecen
Other Study IDs: DE RKEB/IKEB:4364/2015; 094579/2015/OTIG (Other: Health Registration and Training Center Department of Medical Devices)
Record Dates: First submitted 2016-01-13; First posted 2016-01-27 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Cerebral Oxygen Saturation,MCA Velocity,Intraoperative Neurological Symptoms During Carotid Endarterectomy
Keywords: Cerebral oxygen saturation; TCD; NIRS; Carotid endarterectomy
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients without neurological symptoms: carotid endarterectomy patients who dont'have any neurological symptoms after carotid clamping
  Interventions: Device: transcranial Doppler (TCD) and INVOS monitor
- patients with neurological symptoms: carotid endarterectomy patients who have new neurological symptoms after carotid clamping
  Interventions: Device: transcranial Doppler (TCD) and INVOS monitor

INTERVENTIONS:
Device: transcranial Doppler (TCD) and INVOS monitor — Bilateral transcranial Doppler measurements of the blood flow velocity within the middle cerebral arteries: 1. before local anesthesia, 2. after the onset of local anesthetic, but before skin incision, 3. intraoperatively before clamping the internal carotid artery, 4. one minute after clamping the internal carotid artery, 5. five minutes after clamping the internal carotid artery, 6. fifteen minutes after clamping the internal carotid artery, 7. directly after the restoration of blood flow in the internal carotid artery, 8. postoperatively, 4-6 hours after the intervention.

SUMMARY:
The primary endpoint of our study is to determine whether neurological symptoms (aphasia, paresis, loss of consciousness, numbness) occur after clamping the internal carotid artery, and if so, changes showed by transcranial Doppler or INVOS monitor is more sensitive regarding the symptoms? Secondary endpoint: the degree of change in the measured parameters after the internal carotid artery is clamped, and if there is any difference between the operated and non-operated sides?

DETAILED DESCRIPTION:
Investigation of blood flow velocity in the middle cerebral artery and oxygen saturation of the brain bilaterally during carotid endarterectomy carried out in local anesthesia in patients with and without neurological symptoms using transcranial Doppler (TCD) and INVOS monitor.

Zoltán Gyöngyösi Study protocol

The primary endpoint of our study is to determine whether neurological symptoms (aphasia, paresis, loss of consciousness, numbness) occur after clamping the internal carotid artery, and if so, changes showed by transcranial Doppler or INVOS monitor is more sensitive regarding the symptoms? Secondary endpoint: the degree of change in the measured parameters after the internal carotid artery is clamped, and if there is any difference between the operated and non-operated sides?

Patients and Methods

Outpatient examination, preparation and anesthesia of the patients:

* ECG test
* Echocardiography, if it is necessary due to the cardial status of the patient.
* Indication of surgical intervention provided by the cerebrovascular outpatient clinic, with attached carotid ultrasound and angiography results.

Surgical anesthesia:

* Superficial and deep cervical block with 3.75% ropivacaine (50ml ropivacaine 3.75%) (incase of allergy bupivacaine should be used)
* Securing venous catheter, infusion of Lactated-Ringer or Voluven solution.
* In case of pain topical administration of Lidocaine by the surgeon, intravenous administration of 25-50ug Fentanyl or 1 vial of Algopyrin.

Intraoperative measurements:

* Bilateral transcranial Doppler measurements of the blood flow velocity within the middle cerebral arteries: 1. before local anesthesia, 2. after the onset of local anesthetic, but before skin incision, 3. intraoperatively before clamping the internal carotid artery, 4. one minute after clamping the internal carotid artery, 5. five minutes after clamping the internal carotid artery, 6. fifteen minutes after clamping the internal carotid artery, 7. directly after the restoration of blood flow in the internal carotid artery, 8. postoperatively, 4-6 hours after the intervention.
* Recording mean arterial pressure with each TCD measurement.
* Recording cerebral saturation (INVOS) with each TCD measurement.
* Recording any anti-hypertensive therapy in the postoperative phase.
* Recording heart rate.
* Recording arterial oxygen saturation.
* Recording the patients' neurological status with each TCD measurement and continuous neurological monitoring while the internal carotid artery is clamped.

ELIGIBILITY:
Inclusion Criteria:

* 100 patients awaiting carotid artery endarterectomy carried out in regional anesthesia.
* Age: patients over 18 years.
* Gender: both female and male patients are included in the study.
* Medical equipment: venous catheter, arterial catheter for invasive blood pressure monitoring.
* Bilateral continuous measurement of the middle cerebral arteries with Transcranial Doppler.
* Bilateral continuous measurement of the cerebral saturation with INVOS monitor.

Exclusion Criteria:

* Allergy to ropivacaine, bupivacaine.
* Patients who does not consent to the awake surgery or does not sign the informed consent of the study.
* If the patient is either psychologically or neurologically unsuitable for the awake surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 100 patients awaiting carotid artery endarterectomy carried out in regional anesthesia.
  * Age: patients over 18 years.
  * Gender: both female and male patients are included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
to determine the changes in MCA flow velocity in patient with intraoperative neurological symptoms | 15 month
  (aphasia, paresis, loss of consciousness, numbness) occur after clamping the internal carotid artery, and if so, to determine the changes in MCA flow velocity in patient with intraoperative neurological symptoms
  Recording mean arterial flow velocity with each TCD measurement.
to determine the changes in cerebral O2 saturation in patient with intraoperative neurological symptoms | 15 month
  Recording cerebral saturation (INVOS) with each measurement.

SECONDARY OUTCOMES:
the degree of change in the measured parameters during clamp and declamp after the internal carotid artery is clamped, if there is any difference between the operated and non-operated sides? | 15 month
  Recording mean arterial pressure with each TCD measurement. Recording cerebral saturation (INVOS) with each measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Béla Fülesdi, MD,PhD,DSci, Principal Investigator — Hungary University of Debrecen Debrecen, Hungary, 4032
Locations (2):
- Hungary (2):
  - University of Debrecen, Debrecen, Hajdú-Bihar
  - University of Debrecen, Debrecen

REFERENCES:
- [Result] Williams IM, Mead G, Picton AJ, Farrell A, Mortimer AJ, McCollum CN. The influence of contralateral carotid stenosis and occlusion on cerebral oxygen saturation during carotid artery surgery. Eur J Vasc Endovasc Surg. 1995 Aug;10(2):198-206. doi: 10.1016/s1078-5884(05)80112-1. PMID 7655972
- [Result] Pennekamp CW, Immink RV, den Ruijter HM, Kappelle LJ, Bots ML, Buhre WF, Moll FL, de Borst GJ. Near-infrared spectroscopy to indicate selective shunt use during carotid endarterectomy. Eur J Vasc Endovasc Surg. 2013 Oct;46(4):397-403. doi: 10.1016/j.ejvs.2013.07.007. Epub 2013 Aug 21. PMID 23973277